CLINICAL TRIAL: NCT04144166
Title: Evaluation of Capillary Refill Index
Acronym: CRI
Status: Completed | Type: Observational
Sponsor: Nihon Kohden (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-011-004
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Perfusion; Complications
Keywords: capillary refill time; peripheral perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: capillary refill index (CRI) — a waveform analysis method using a pulse oximeter to assess peripheral perfusion

SUMMARY:
Comparison of a peripheral perfusion assessment method using a pulse oximeter to the conventional capillary refill time visually assessed by a clinician.

DETAILED DESCRIPTION:
A new technology, capillary refill index (CRI), to assess peripheral perfusion status quantitatively using pulse oximeter waveforms is being developed. The conventional capillary refill time (CRT) is widely used in clinical settings as a gold standard to assess peripheral perfusion.

The objective of this study is to evaluate the capability of CRI to predict altered peripheral perfusion determined with the conventional CRT test. Predictive capability of CRI needs to be assessed to achieve a goal to provide clinicians with an alternative method to the conventional CRT.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 18 years of age or older
2. Patients who present to the ED or who are admitted to the ICU of North Shore University Hospital (NSUH)

Exclusion Criteria:

1. Pregnant
2. Prisoners
3. Finger, hand or forearm anatomical anomaly or disease that may interfere with attaching a pulse oximeter sensor
4. Patients' deemed clinically unstable by the clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults in ED or admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timmy Li, PhD, Principal Investigator — Admin Dir Clinical Research Emergency Medicine, Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: Adult emergency department (ED) patients, both males and females without regards to ethnic and racial backgrounds. CRT and CRI measurements were conducted with following methods for each subject in a relaxed position (seated or lying down) with relaxed hands. The subject's most accessible hand (right or left) was used. Each measurement of visual CRT and device CRI were performed alternately and were repeated three times each for a total of six compressions per subject.
  Visual CRT measurement using a stopwatch An investigator (an ED physician) compressed the fingertip of the subject's index or middle finger for five seconds, signaled by "start compression" and "release compression" beep sounds. When the fingertip was released from the compression, the investigator began the visual CRT measurement. The investigator held a stopwatch in the hand that did not perform the compression and used this stopwatch to measure CRT.
  CRI measurement by the investigational device The SpO2 sensor probe was applied to either the index or middle fingertip of the same hand of the subject used in the CRT measurement, depending upon which fingertip was compressed in the CRT measurement. The investigator who measured the visual CRT was blinded from the measured value of the CRI measurement.
Period: Overall Study
Arm/Group | All Subjects
Started | 60
Completed | 57
Not Completed | 3
Not completed — Discharged before study start | 1
Not completed — Pregnancy | 1
Not completed — Nail polish could not be removed from finger | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 57
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49.0 [38.0 to 66.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32
  Black or African American | 8
  Asian | 3
  Other/Multiracial | 13
  No designation | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57
Fitzpatrick Skin Tone Scale [Number; unit: participants] — Fitzpatrick skin tone scale is a numerical classification schema for human skin color. The scales range from 1 - fairest skin to 6 - very dark pigment skin. A visual chart comparison was used for assignment of each subject. Results (see later) only addressed a comparison of subjects in Fitzpatrick 1, 2 or 3 versus subjects in Fitzpatrick 4, 5 of 6.
  participants
    Fitzpatrick skin tone - 1 | 9
    Fitzpatrick skin tone - 2 | 13
    Fitzpatrick skin tone - 3 | 14
    Fitzpatrick skin tone - 4 | 7
    Fitzpatrick skin tone - 5 | 7
    Fitzpatrick skin tone - 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Predictive Capability of the Altered Peripheral Perfusion
Description: The area under the curve (AUC) of the receiver operator characteristic (ROC) curve analysis on CRI values to predict probability of altered peripheral perfusion determined with the CRT test.
Time Frame: < 30 min *right after enrollment
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Sensitivity and Specificity to Predict Low Peripheral Perfusion: Ability to differentiate altered peripheral perfusion with a CRI cutoff value of 3.37 s for low CRT (> 2 s) and very low CRT (> 3 s)
Arm/Group | Sensitivity and Specificity to Predict Low Peripheral Perfusion
Number analyzed (Participants) | 57
probability
  Optimal CRI (3.37 s) low peripheral perfusion sensitivity | 0.89 [0.71 to 0.98]
  Optimal CRI (3.37 s) low peripheral perfusion specificity | 1.00 [0.88 to 1.00]
  Optimal CRI (3.37 s) very low peripheral perfusion sensitivity | 0.94 [0.73 to 1.00]
  Optimal CRI (3.37 s) very low peripheral perfusion specificity | 0.82 [0.67 to 0.93]
  AUC low peripheral perfusion (> 2 s) | 0.986 [0.944 to 0.997]
  AUC very low peripheral perfusion (> 3 s) | 0.910 [0.807 to 0.960]

2. Secondary Outcome: Correlation of Device CRI to Conventional (Visual) CRT
Description: Spearman's correlation coefficient to assess the correlation between CRI and CRT values.
Time Frame: < 30 min *right after enrollment
Measure: Number (95% Confidence Interval); unit: Spearman's correlation coefficient
Groups:
- Correlation Between CRI and CRT Values: Spearman's correlation method to determine relationship between median device CRI and median device CRT measurements.
Arm/Group | Correlation Between CRI and CRT Values
Number analyzed (Participants) | 57
Spearman's correlation coefficient | 0.866 [0.782 to 0.919]
Statistical Analysis 1: Comparison: Correlation Between CRI and CRT Values; Mean value for visual CRT and median value for device CRI were calculated for each participant. 3 values were measured (each) for CRT and CRI. Mean value is equal to SUM(m1,m2,m3)/3. Median value was then calculated for the set (57) of calculated mean visual CRT and mean device CRI. Median value is equal to the middle value of the series of mean values. All measurements are in units of seconds; Test type: Other; See above; See above

3. Post Hoc Outcome: Independence of Age Impact on CRI Measurement for Low Peripheral Perfusion (CRT > 2 Seconds)
Description: Demonstrate that age is not a variant for CRI measurement
Time Frame: < 30 min *right after enrollment
Population: Patients < 60 years vs. >= 60 years
Measure: Number (95% Confidence Interval); unit: probabllity
Groups:
- All Subject >= 60 Years: All subject >= 60 years
- All Subjects < 60 Years: All subjects < 60 years
Arm/Group | All Subject >= 60 Years | All Subjects < 60 Years
Number analyzed (Participants) | 23 | 34
probabllity | 0.992 [0.888 to 1.000] | 0.982 [0.901 to 1.000]

4. Post Hoc Outcome: Independence of Fitzpatrick Skin Tone Score on CRI Measurement for Low Peripheral Perfusion (CRT > 2 Seconds)
Description: Demonstrate that skin tone is not a variant for CRI measurement
Time Frame: < 30 min *right after enrollment
Population: Subjects with Fitzpatrick skin tone score of 1, 2 or 3 vs. scores of 4, 5, or 6
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- All Subjects With Fitzpatrick Skin Tone Score of 1, 2 or 3: All subjects with FItzpatrick skin tone score of 1, 2 or 3
- All Subjects With Fitzpatrick Skin Tone Score of 4, 5 or 6: All subjects with FItzpatrick skin tone score of 4, 5 or 6
Arm/Group | All Subjects With Fitzpatrick Skin Tone Score of 1, 2 or 3 | All Subjects With Fitzpatrick Skin Tone Score of 4, 5 or 6
Number analyzed (Participants) | 36 | 21
probability | 0.994 [0.993 to 1.00] | 0.981 [0.820 to 0.998]

ADVERSE EVENTS:
Time Frame: 30 min
Description: All adverse events (all cause mortality, serious-adverse, other - not serious) reported to P.I. in written form via data collection form
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

LIMITATIONS AND CAVEATS:
Sample size: Number of required sample size was 54. Detail of the sample size calculation is described in the clinical protocol document. Actual results were 57 subjects, so results are statistically valid with respect to sample size.

Participant flow: Subject discovered to be pregnant and removed from study. Since study is non-invasive and minimal risk, subject and fetus were not exposed to any additional risks. Hospital IRB was notified of deviation and did not require other reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT04144166/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT04144166/ICF_001.pdf